CLINICAL TRIAL: NCT06987253
Title: Assessment of the Efficacy and Safety of OROXID® Oral Solution in Patients With Oral Cavity Surgery
Acronym: OroxSurge
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ENIKAM d.o.o. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OROXID-PR-01-25
Record Dates: First submitted 2025-05-08; First posted 2025-05-23 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Tooth Extrusion; Wound Healing
Keywords: Oral cavity wound; Hydrogen peroxide; Mouthwash
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OROXID® forte (Experimental): Medical device: OROXID® forte oral solution
  Interventions: Device: OROXID® forte oral solution
- Standard of care (Other): Oral solutions are not allowed
  Interventions: Other: Standard of Care (SOC)

INTERVENTIONS:
Device: OROXID® forte oral solution — Patients will use OROXID® forte oral solution two to three times daily for 14 days as an adjunct to standard care.
  Arms: OROXID® forte
Other: Standard of Care (SOC) — Patients will receive standard of care meaning proper tooth brushing without the use of any mouthwash or other products aimed at reducing bacteria in the oral cavity.
  Arms: Standard of care

SUMMARY:
Oral tissue healing is significantly affected by the high bacterial load and constant mechanical stress within the oral cavity. To control bacterial colonization and support healing, both topical and systemic treatments-such as antibiotics and anti-inflammatory agents-are commonly recommended. In addition to pharmacological therapies, mouthwashes containing peroxide, hyaluronic acid, chitosan, or chlorhexidine are often used to maintain low levels of pathogenic bacteria.

However, current recommendations for mouthwash use are primarily based on their antibacterial properties in a healthy oral environment. Evidence supporting their role in promoting wound healing, particularly after oral surgery, remains limited.

OROXID® mouthwash is a medical device formulated with active oxygen (peroxide compounds). It supports the prevention and relief of inflammation in gingival and paranasal tissues through mechanical action: the release of oxygen bubbles helps cleanse tissues by removing debris. OROXID® acts locally on the mucosal microenvironment by moistening, oxygenating, and clearing away particles and dead cells. Additionally, its slightly acidic pH (between 3 and 5) helps inhibit microbial growth.

The investigators hypothesize that OROXID® may reduce post-operative side effects and complications following wisdom tooth extraction and contribute to faster wound healing.

ELIGIBILITY:
Inclusion Criteria:

1. Systemically healthy individuals aged 18 years or older.
2. Indicated for surgical removal of an erupted or unerupted tooth and/or apicoectomy.
3. Ability and willingness to comply with post-operative oral hygiene instructions.
4. Signed informed consent form prior to participation in the study.

Exclusion Criteria:

1. Receipt of periodontal treatment within the past 3 months.
2. Use of mouthwashes or oral gels in the past month.
3. Presence of active gingivitis around the tooth scheduled for extraction.
4. Known allergy to any ingredients of the investigational products.
5. Presence of inflammatory conditions in the oral cavity, such as lichen planus, bullous lesions, or active gingivitis.
6. Immunocompromised individuals.
7. Known allergy to penicillin or diclofenac.
8. Pregnant or breastfeeding women.
9. Smokers who consume more than 15 cigarettes per day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-06 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Modified Landry Index | 7 days
  Differences in the total score of the individual components of the Modified Landry Index between the active and control groups. This entails evaluating the following parameters in a comparative manner using a dichotomic score: gingival color (0 = red, 1 = pink); granulation tissue (0 = present, 1 = absent); tissue epithelialization (0 = partial/1 = complete); swelling (0 = pres- ence, 1 = absent); bleeding on palpation (0 = present, 1 = absent); sup- puration on palpation (0 = present, 1 = absent). The total score, ranging from 0 to 6, reflects the overall quality of healing, with higher scores indicating more favorable outcomes.

SECONDARY OUTCOMES:
Completely Healed Wounds | 14 days
  Proportion of completely healed wounds at 14 days in the active versus control group.
Mean Early Healing Index | 7 and 14 days
  Mean Early Healing Index (EHI) scores will be used to compare the groups. The EHI evaluates key clinical indicators of wound healing, including redness, swelling, bleeding, and epithelialization. Scores range from 0 to 5, with 0 representing very poor healing and 5 indicating excellent healing. Higher EHI scores correspond to more favorable healing outcomes.
Plaque Index | 7 and 14 days
  Differences in Plaque Index (PI) scores between the active and control groups will be evaluated using the Silness and Löe Plaque Index. This index assesses the thickness of dental plaque along the gingival margin based on the following scoring criteria: Score 0 = No plaque score; 1 = Mild plaque along the gingival margin; Score 2 =Moderate layer of plaque along gingival margin, interdental spaces free; Score 3 = Abundant plaque along the gingival margin, interdental spaces filled with plaque. Higher scores indicate poorer oral hygiene and greater plaque accumulation.
Pain Relief | In the first 7 days
  Assessment of additional analgesic use (measured in days) will be conducted to compare the active and control groups.
Infection rate | 7 and 14 days
  Incidence of post-operative infections in each group

CONTACTS AND LOCATIONS:
Overall Officials: Tadej Dovšak, PhD, Principal Investigator — Krizaj d.o.o.
Locations (1):
- Klinika Križaj, Muljava, Občina Ivančna Gorica, Slovenia

IPD SHARING:
Plan to Share IPD: No
As a company operating under the jurisdiction of the EU, the organization is subject to the General Data Protection Regulation (GDPR), which imposes strict requirements on the processing and sharing of personal data, including health-related information. Individual Participant Data (IPD) from clinical trials is considered sensitive personal data under GDPR.
  Even when data is anonymized or pseudonymized, sharing IPD with third parties-especially outside the EU-requires careful assessment of data protection safeguards, appropriate legal basis, and in some cases, additional participant consent. Unless all conditions for lawful data transfer and processing are met, including compliance with GDPR Articles 44-50 concerning international data transfers, the sharing of IPD is not permitted.
  For this reason, and to ensure full compliance with EU data protection regulations while safeguarding the privacy and rights of study participants, individual-level data cannot currently be shared.